CLINICAL TRIAL: NCT04269018
Title: The Effect of Mobile Text Message on Behavioral Risks of Cancer Among College Students, Northeast Ethiopia: A Randomized Controlled Trial
Brief Title: The Effect of Mobile Text Message on Behavioral Risks of Cancer: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Foziya Mohammed Hussien, lecturer, Wollo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24
Record Dates: First submitted 2020-02-09; First posted 2020-02-13 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Behavioral Risks of Cancer

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to intervention and control group, the intervention group will be received daily text message while the controls will receive general health messages once a week.
Who Masked: Participant
Masking Description: To maintain blinding, randomization will occur after the baseline assessment and both groups will receive welcome message for participating in the study. Then motivational and general healthy related texts will be delivered to controls one times per week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer specific Mobile text message (Experimental): This arm will receive daily mobile text message related with cancer risks and prevention
  Interventions: Behavioral: Cancer specific Mobile text message
- general health messages (Active Comparator): This arm will receive general health message once a week
  Interventions: Behavioral: General health messages

INTERVENTIONS:
Behavioral: Cancer specific Mobile text message — The intervention is cancer specific lifestyle mobile text messages daily for 2 months
  Arms: Cancer specific Mobile text message
Behavioral: General health messages — Daily text related with general health message
  Arms: general health messages

SUMMARY:
Summary Background: Cancer is a public health problem in Ethiopia. A third of cancer deaths are preventable. Its effects can be significantly reduced if effective interventions are put in place to control risk factors. Text-messaging has been currently targeted as a simple tool for providing people with health information. Thus this study aimed to measure the effectiveness of text message in behavioral risk factors that is helpful to raise cancer awareness and promote cancer prevention and control in this country.

Methods: A randomized control trial will be used to measure the effectiveness of mobile text message in behavioral risk factor of cancer among Governmental Collage students in Dessie City and utilize quantitative method of data collection. Data will be collected on a total of 80 intervention and 80 controls using structured questionnaire. Socio-demographic, health belief variables and behavioral risk factor of cancer will be collected before and after intervention. Text message will be provided based on health belief model. Data will be entered using Epidata version 3.1 and will be exported to STATA version 13.0 for cleaning and analysis. Liner regression will be applied to identify predictors of behavioral risk factor of cancer. Student's paired samples t-test will be used to test changes in terms of HBM variables and behavioural outcomes. Analysis of Covariance will be used to test over group comparison.

DETAILED DESCRIPTION:
The study will be a single blind randomized controlled trial, which utilize quantitative method of data collection. College students who will receive a mobile text message about the behavioral risks of cancer and prevention mechanism will be considered as intervention groups while controls will be those who receive a text message related with general health once a week. A total of 160 (80 interventions and 80 controls) students will be included in the study using simple random sampling technique. After the baseline assessment, participants will be randomized to either usual care (control) or the text message intervention group in a uniform 1:1 (control: intervention) allocation ratio, using computer-based randomization service.

Self-administered questionnaire will be used to assess baseline and end line data of behavioral risk factors and other variables. Participants in the control group will receive an initial text message welcoming them to the study, but they will not receive the text message support program. The intervention group will receive a text message support program, where they will receive seven messages per week at random times and days for two months. The text message will be prepared and delivered based on health belief model (HBM), the items of this subscale will be measured on a Likert scale ranging from 1= "Strongly disagree" to 5 = "Strongly agree". Tobacco use, harmful use of alcohol, unhealthy diet and physical inactivity with a series of items will be used to measure the behavioral outcomes the items in this subscale will be measured on a Likert scale.

Validity of the items will be measured by an expert panel of specialists in health education and nutrition. They will judge about the necessity and relevance of the scale items. To control the data quality all data collectors will be trained for two days. Supervisors will monitor data collection process and the principal investigator will visit frequently. The questionnaire will be first prepared in English language and translated to Amharic and again re-translated in to English by another person to check for consistency. About 10% of the questionnaire will be pretested and internal consistency will be checked. Completeness of the collected data will be checked during data collection.

The data will be checked for completeness and consistency, then categorized, coded and entered using Epidata version 3.1 to minimize error. Then, the clean data will be exported to Stata version 14 for analysis. Normality of the data will be checked through Kolmogorov-Smirnov test. Student's paired samples t-test will be used to test within-group changes in terms of health belief model (HBM) variables and behavioral outcomes. The analysis of Covariance will be used to make over-group comparisons. Data will be reported as mean ± standard deviation. The significance level for all of the results will be presented at the P<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* College students aged 18 to 35

Exclusion Criteria:

* Mental and physical disability, those who already have diagnosed cancer

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | on average 6 months
  For measuring physical activity International Physical Activity Questionnaires (IPAQ) will be used. The questions will ask the time study participants spent being physically active in the last 7 days. Then, it will be summarized as Metabolic Equivalents (METs).
Health dietary score | on average 6 months
  Healthy diet score will be assessed the health diet score adapted from the WHO list of healthy diet foods, which is a Likert scale ranged from 1 to 6.
Tobacco use | on average 6 months
  Tobacco smoking will be assessed using a series of questions adopted from the World Health Organization (WHO), which used to assess the duration, quantity and frequency of smoking within one month.
Alcohol intake | on average 6 months
  Alcohol consumption will be assessed using a tool adopted from National Institute on Alcohol Abuse and Alcoholism (NIAAA), which used to assess participants consumption in the past 1 month.
Risk perception | on average 6 months
  Risk perception will be measured using health belief model variables: perceived susceptibility towards cancer, perceived severity of cancer, perceived benefits of adopting behaviors, perceived barriers to adopting behaviors, perceived self-efficacy for adopting dietary behaviors and internal cues for adopting dietary behaviors, the items of this subscale will be measured on a Likert scale ranging from 1= "Strongly disagree" to 5 = "Strongly agree".

REFERENCES:
- [Derived] Hussien FM, Hassen AM, Asfaw ZA, Ahmed AY, Dawed YA, Asfaw AH, Amsalu ET, Hassen HY. Knowledge and practice regarding the behavioural risks of cancer among college students in Ethiopia. Ecancermedicalscience. 2022 Jan 13;16:1343. doi: 10.3332/ecancer.2022.1343. eCollection 2022. PMID 35242224
- [Derived] Hussien FM, Hassen AM, Asfaw ZA, Ahmed AY, Hassen HY. The effect of mobile text messages on knowledge and perception towards cancer and behavioral risks among college students, Northeast Ethiopia: A randomized controlled trial protocol. PLoS One. 2021 Jul 9;16(7):e0253839. doi: 10.1371/journal.pone.0253839. eCollection 2021. PMID 34242256